CLINICAL TRIAL: NCT02151305
Title: The Influence of Propofol and Sevoflurane on Hemostasis During Ophthalmic Surgery: Rotational Thromboelastographic Study.
Brief Title: Different Hemostasis According to the Anesthetic Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Pf, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ROTEM_anesthesia
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Cataract; Retina Detachment; Pterygium; Keratitis; Vitreous Hemorrhage
MeSH Terms: conditions — Cataract; Retinal Detachment; Pterygium; Keratitis; Vitreous Hemorrhage | interventions — Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Total intravenous anesthesia group (Experimental): This group received propofol and remifentanil for the maintenance of general anesthesia.
  Interventions: Drug: Propofol, remifentanil
- Inhalation anesthesia group (Experimental): This group received sevoflurane for the maintenance of general anesthesia.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol, remifentanil
  Arms: Total intravenous anesthesia group
Drug: Sevoflurane
  Arms: Inhalation anesthesia group

SUMMARY:
We investigated the hemostatic differences according to the main anesthetic agents by analyzing rotational thromboelastometry (ROTEM) under the hypothesis that propofol-based anesthesia would impair postoperative coagulability more than the sevoflurane-based anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All patient scheduled for ophthalmic surgery under general anesthesia
* American Society of Anesthesiologist physical status I or II

Exclusion Criteria:

* hematologic disorder
* severe anemia
* liver disease
* kidney disease
* taking a medication interfering with hemostasis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Clotting time of ROTEM | 10 minutes before the induction of anesthesia, 1 h after finishing anesthesia
Clot firmness time of ROTEM | 10 minutes before the induction of anesthesia, 1 h after finishing anesthesia
Alpha angle of ROTEM | 10 minutes before the induction of anesthesia, 1 h after finishing anesthesia
Maximum clot firmness of ROTEM | 10 minutes before the induction of anesthesia, 1 h after finishing anesthesia

SECONDARY OUTCOMES:
Hemoglobin | 10 minutes before the induction of anesthesia
Hematocrit | 10 minutes before the induction of anesthesia
Platelet count | 10 minutes before the induction of anesthesia
International normalized ratio of prothrombin time | 10 minutes before the induction of anesthesia
Activated partial thromboplastin time | 10 minutes before the induction of anesthesia
Fibrinogen | 10 minutes before the induction of anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea